CLINICAL TRIAL: NCT01366742
Title: Natural History of Human Papillomavirus From Infection to Neoplasia in Adolescents and Young Women - Effect of Tobacco on Cervical Neoplasia in Young Women
Brief Title: Natural History of HPV From Infection to Neoplasia in Adolescents and Young Women
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11-05580; R37CA051323 (NIH)
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Human Papillomavirus; CIN 2; CIN 3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Rbc, WBC vaginal lavages ,cytology,saliva ,anal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HPV Cohort: Sexually active young women aged 12 to 22 years of age without a previous history of CIN. Women are not eligible for entry if pregnant or known immunosuppression.

SUMMARY:
The natural history of human papillomavirus (HPV) is most likely influenced by both innate and adaptive mucosal immunity. More specifically, we hypothesize that Toll like receptors (TLR) play an important role in cervical innate immunity to HPV through secretions of proinflammatory, chemotactic and anti-viral cytokines. Up-regulated TLR expression will also result in activation of dendritic cells and T cells that in turn will promote a T helper (Th) l like response through secretion of several cytokines and consequently, the induction of a successful cell mediated immune (CMI) response.

DETAILED DESCRIPTION:
The natural history of HPV is most likely influenced by both innate and adaptive mucosal immunity. More specifically, we hypothesize that Toll like receptors (TLRs) play an important role in cervical innate immunity to HPV through secretions of proinflammatory, chemotactic and anti-viral cytokines. Up-regulated TLR expression will also result in activation of dendritic cells and T cells that in turn will promote a Thl like response through secretion of several cytokines and consequently, the induction of a successful cell mediated immune (CMI) response.

We propose to: 1) examine, in cervical cell samples, the association among TRL expression, TRL-associated cytokines that mediate innate immunity and clearance of incident HPV infection; 2) examine, in cervical cell samples, the association among TRL expression, TRL-associated cytokines that induce and mediate adaptive immunity and HPV clearance; and 3) examine the association among TLR induced Th-1 responses measured in cervical cell samples, HPV specific CMI responses detected in peripheral blood (PB) and HPV clearance. Adolescent and young women who were a) entered into the cohort during the initial 1990-1995 period and have continued to be followed and b) entered into the cohort during the last recruitment wave (2000-2005) will be asked to continue followup for an additional five years (2005-2010). These women will have been well characterized at the time of the initiation of this study with HPV at their entry visit and 4-month interval sampling for HPV DNA, cytology, bacterial vaginosis, colpophotographs (assessment of cervical maturation), C. trachomatis and N. gonorrhea testing, cervical cell cytokines by reverse transcriptase polymerase chain reaction (RT-PCR) and peripheral blood (PB) CMI for HPV 16 positive women. Women will be continued to be characterized for the above at the same intervals through-out the follow-up. Measures of innate and adaptive immunity by RT PCR using cervical cells and by Luminex technology have been added to the same 4 month interval testing as HPV DNA, cytology and other cervical cytokines described. Women positive for HPV 16 will get additional blood for CMI using Interferon (IFN)-y Enzyme linked immunospot (EliSpot) technique for detection of anti-E6 and E7 responses. We also examine the natural history of anal HPV in these women. We acknowledge that this design simplifies the pleiotropic nature of cytokines. However, we feel that this model reflects plausible mechanisms involved in HPV control and is feasible to test in our cohort. Information garnered from this type of study will be critical in developing vaccine strategies and therapies as well as illuminating immune responses developed in the mucosal epithelium.

ELIGIBILITY:
Inclusion:

* Age 12 to 22 years
* Sexually active less than 6 years
* Received one dose of the HPV vaccine

Exclusion:

* Planning on moving in 3 years
* Prior history of treatment for CIN
* Immunocompromised (ie transplant patient, HIV)
* Pregnant

Ages: 13 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 1987-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Cervical Intraepithelial neoplasia (CIN) 2/3 | 1990 to current
  Observational study of women with HPV

SECONDARY OUTCOMES:
HPV persistence | 1990 to present
  observational study of women with HPV

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Barbara Moscicki, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - SFSU Student Health Center, San Francisco, California
  - HPV Study - San Leandro Office, San Leandro, California